CLINICAL TRIAL: NCT03358095
Title: Cancer of the Head of the Pancreas: Early Surgery or Preoperative Biliary Drainage? A Prospective Study
Brief Title: Cancer of the Head of the Pancreas: Early Surgery or Preoperative Biliary Drainage?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators busy with other projects at the moment.
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, Head of department, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early surgery vs PBD
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer; Biliary Stasis
MeSH Terms: conditions — Pancreatic Neoplasms; Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (No Intervention): Patients in this group proceed to pancreatic resection within 2 week of recruitment.
- Preoperative biliary drainage (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) is used to place an endoprosthesis to the biliary ducts to drain biliary stasis, and the patients proceed to pancreatic resection within 6 weeks of recruitment.
  Interventions: Device: Tannenbaum Fr 10 stent or WallFlex stent

INTERVENTIONS:
Device: Tannenbaum Fr 10 stent or WallFlex stent — A plastic or metallic endoprosthesis is placed to the biliary ducts.
  Arms: Preoperative biliary drainage

SUMMARY:
Surgical resection is the only option for cure for patients with a resectable tumor located at the head of the pancreas. At the time of diagnosis, these patients often suffer from jaundice. Studies have suggested, that jaundice might increase the risk of developing a serious postoperative complication. Preoperative biliary drainage is widely used, because it is considered to improve the surgical outcome and reduce the amount of postoperative complications. There are also studies that suggest the opposite. In these studies the overall complication rate with patients who underwent preoperative biliary drainage was higher than in the patients who were operated right away. A significant amount of these complications were related to the biliary drainage process itself. However, preoperative biliary decompression is widely used in many centers as many surgical centers don't possess the needed resources to arrange early surgery. The benefits and risks of this procedure remain unclear. This multicenter trial aims to compare the surgical outcome and the rate of serious complications in patients who proceed directly to early surgery and patients who have preoperative biliary drainage.

ELIGIBILITY:
Inclusion Criteria:

* Patients in this study must have a resectable tumor of the head of the pancreas, and no evidence of distant metastasis or local vascular involvement. At the beginning of the study it's not necessary to have an accurate histologic diagnosis, the tumor might be malignant or benign. The patients also have jaundice with a total serum bilirubin level of 40-250µmol/l, and are fit enough to be considered for an early surgery.

Exclusion Criteria:

* Patients with ongoing cholangitis, neoadjuvant treatments or previous biliary drainage with stenting by means of ERCP or PTC (Percutaneous Transhepatic Cholangiogram) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emerged complications related to surgery or preoperative endoscopy within 120 days of surgery | 120 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sini Vehviläinen, MD, Study Chair — Helsinki University Central Hospital; Hanna Seppänen, MD, PhD, Study Chair — Helsinki University Central Hospital; Arto Kokkola, MD, PhD, Study Chair — Helsinki University Central Hospital; Marianne Udd, MD, PhD, Study Chair — Helsinki University Central Hospital; Outi Lindström, MD, PhD, Study Chair — Helsinki University Central Hospital; Johanna Louhimo, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Gaag NA, Kloek JJ, de Castro SM, Busch OR, van Gulik TM, Gouma DJ. Preoperative biliary drainage in patients with obstructive jaundice: history and current status. J Gastrointest Surg. 2009 Apr;13(4):814-20. doi: 10.1007/s11605-008-0618-4. Epub 2008 Aug 23. PMID 18726134
- [Background] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702